CLINICAL TRIAL: NCT01584895
Title: Cardiac Rehabilitation in Patients With Continuous Flow Left Ventricular Assist Devices:Rehab VAD Trial
Acronym: RehabVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Dennis J. Kerrigan, Senior Exercise Physiologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: hfhs-pc-RehabVAD
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehab (Experimental): Patients randomized into early cardiac rehabilitation
  Interventions: Behavioral: Cardiac Rehabilitation
- Control (No Intervention): No cardiac rehabilitation until after 6 week post assessment.

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — A standard cardiac rehabilitation program consisting of 3 days per week of supervised exercise and education.
  Arms: Rehab

SUMMARY:
Cardiac rehabilitation programs improve mortality, functional capacity, and quality of life, for a variety of patients with heart disease. It stands to reason that patients with LVADs might therefore also benefit from the same structured exercise training, education, and clinical surveillance. One potential benefit of cardiac rehabilitation in this patient population is reversal of the skeletal muscle atrophy that occurs due to extended periods of poor peripheral perfusion (i.e. before implantation) and prolonged sedentary behavior.

Purpose: The purpose of this proposed study is to examine the effects of a 6-week exercise program on cardiorespiratory fitness, quality of life, and device flow rate in patients with recently implanted LVADs.

Methods: 30 patients with recently implanted LVADs will be referred by the Henry Ford Hospital Advanced Heart Failure Program once the patient is deemed appropriate for exercise. Before enrollment into cardiac rehabilitation patients will undergo a six minute walk test and graded exercise stress test on a treadmill to determine exercise capacity. Additionally, a quality of life questionnaire will be given.

Following the stress test, patients will be randomized (2 to 1 ratio) into either cardiac rehabilitation or control. Those chosen to be in the control group will be encouraged to maintain daily activities; those in the rehabilitation group will partake in 6 weeks of a standard cardiac rehabilitation program. This will consist of 3 days a week of supervised exercise as well as education regarding diet and lifestyle modifications.

At 6 weeks after randomization both groups will again undergo fitness assessments and retake the quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Continuous flow left ventricular assist device
* Implanted within the past six months
* Approval from cardiologist to participate in cardiac rehabilitation
* Age greater or equal to 18 years
* No history of cardiac rehabilitation participation since receiving a LVAD

Exclusion Criteria:

* Orthopedic limitations to perform exercise
* Current infection related to LVAD
* Severe anemia
* Recent CVA related to LVAD implant that affects ability to exercise
* Unable to attend cardiac rehabilitation at Henry Ford Hospital
* Uncontrolled metabolic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary fitness | six weeks
  Peak VO2 as measured on a treadmill using gas exchange

SECONDARY OUTCOMES:
Quality of life | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Kerrigan, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- William Clay Ford Center for Athletic Medicine, Detroit, Michigan, United States

REFERENCES:
- [Background] Kerrigan DJ, Williams CT, Ehrman JK, Bronsteen K, Saval MA, Schairer JR, Swaffer M, Keteyian SJ. Muscular strength and cardiorespiratory fitness are associated with health status in patients with recently implanted continuous-flow LVADs. J Cardiopulm Rehabil Prev. 2013 Nov-Dec;33(6):396-400. doi: 10.1097/HCR.0000000000000024. PMID 24189213
- [Result] Kerrigan DJ, Williams CT, Ehrman JK, Saval MA, Bronsteen K, Schairer JR, Swaffer M, Brawner CA, Lanfear DE, Selektor Y, Velez M, Tita C, Keteyian SJ. Cardiac rehabilitation improves functional capacity and patient-reported health status in patients with continuous-flow left ventricular assist devices: the Rehab-VAD randomized controlled trial. JACC Heart Fail. 2014 Dec;2(6):653-9. doi: 10.1016/j.jchf.2014.06.011. Epub 2014 Oct 22. PMID 25447348